CLINICAL TRIAL: NCT07055256
Title: Elucidating the Role of STAT3 in Epithelial-microbiome Interaction During Periodontitis and Peri-implantitis
Acronym: STAT3EpPPi
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/07; 1231350 (Other Grant/Funding Number: FONDECYT regular); 1231728 (Other Grant/Funding Number: FONDECYT regular); 21221003 (Other Grant/Funding Number: ANID doctorado nacional); 22-004 (Other Grant/Funding Number: Osteology Research Scholarship); 22/385 (Other Grant/Funding Number: PIDFU/PRE-PID)
Record Dates: First submitted 2025-06-25; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-04

CONDITIONS: Periodontitis; Peri-implantitis
Keywords: Periodontitis; Peri-implantitis; STAT3; Epithellial cells
MeSH Terms: conditions — Periodontitis; Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Periodontitis and peri-implantitis are highly prevalent immuno-inflammatory pathologies, characterized by a series of intracellular signals, which, as a consequence of the interaction of the gingival epithelium with the dysbiotic microbiome, lead to an exacerbated immuno-inflammatory response, ultimately resulting in tissue loss around teeth and implants. STAT3 is a transcription factor that plays a key role in inflammatory diseases, which when phosphorylated (pSTAT3) promotes the transcription of genes with immuno-defensive functions. STAT3 phosphorylation has only been reported during experimental periodontitis, but our preliminary results reveal a higher number of epithelial cells with the presence of pSTAT3 in subjects with periodontitis. Other studies have reported greater STAT3 activation in oral keratinocyte cells stimulated with LPS from P. gingivalis, which and F. nucleatum are abundant bacterial species in both pathologies. On the other hand, inhibition of the STAT3 pathway is a therapeutic target in multiple inflammatory diseases, where inhibitors such as C188-9 have shown a direct effect on STAT3 signaling. A better understanding of this signaling pathway in periodontitis and peri-implantitis could allow for future complementary therapies for these diseases.

Based on the above, the hypothesis of this project is:

"During periodontitis and peri-implantitis, there is greater activation of STAT3, particularly at the level of the gingival epithelium, inducing an increase in immune-defensive function in response to microbial dysbiosis and specific constituents of the microbiota associated with these pathologies compared to gingival health."

General objective: To evaluate STAT3 activation and its immune-defensive function during gingival health, periodontitis, and peri-implantitis, specifically at the level of the gingival epithelium, in response to microbial dysbiosis and specific bacteria associated with these periodontal conditions.

Objective 1: To characterize STAT3 activation and immune-defensive function in gingival tissue during gingival health, periodontitis, and peri-implantitis. The investigators will obtain gingival tissue samples from the three conditions through a clinical study. These samples will be processed by Western blot and immunofluorescence to determine pSTAT3. In addition, RT-qPCR will determine the expression of genes related to its immune-defensive function.

Objective 2: To determine STAT3 activation and its immune-defensive function in oral keratinocytes in response to the subgingival biofilm associated with gingival health, periodontitis, and peri-implantitis: Subgingival microbiota samples will be obtained from the three conditions, and the microbiome related to each condition will be characterized by massive sequencing of the 16S rDNA gene. Furthermore, through an in vitro study, oral keratinocyte cells will be stimulated with the obtained samples, and the expression of genes related to their immune-defense function will be determined by Western blot, pSTAT3, and RT-qPCR. The effect of STAT3 inhibition using C188-9 will be subsequently evaluated.

Objective 3: Determine STAT3 activation and its immune-defense function in oral keratinocytes in response to specific bacteria associated with gingival health, periodontitis, and peri-implantitis. Through an in vitro study, oral keratinocyte cells will be infected with reference strains of S. sanguinis, P. gingivalis, and F. nucleatum, and the expression of genes related to their immune-defense function will be determined by Western blot, pSTAT3, and RT-qPCR.

The investigators hope to achieve greater activation of STAT3 and increased expression of genes related to the immune-defensive response of the gingival epithelium during periodontitis and peri-implantitis. The investigators also hope to determine the effect of STAT3 inhibition, expecting a reduction in the expression of genes related to this response.

DETAILED DESCRIPTION:
Aim: To characterize STAT3 activation and immune defense function in gingival tissue during gingival health, periodontitis, and peri-implantitis.

Subject Selection:

This study will comply with the Declaration of Helsinki (October 2013) and Chilean legal and regulatory requirements. The study will be conducted at the Dental Clinic of the Faculty of Dentistry of the University of Chile.

Subjects attending the Dental Clinic of the Faculty of Dentistry of the University of Chile and diagnosed with gingival health, periodontitis, and peri-implantitis, according to the classification of periodontal and peri-implant diseases, will be recruited and examined.

All subjects must sign an informed consent form previously validated by an ethics committee and meet the following inclusion and exclusion criteria:

Inclusion Criteria:

Patients in the Gingival Health Group:

1. Meet the case definition of gingival health.
2. ≥18 years of age.
3. Willingness to donate gingival tissue and collect microbiological samples for the study.

Patients in the Periodontitis Group:

1. Meet the case definition of periodontitis.
2. ≥18 years of age.
3. Willingness to donate gingival tissue and collect microbiological samples for the study.

Patients in the Peri-Implantitis Group:

1. Meet the case definition of periodontitis and peri-implantitis.
2. ≥ 18 years of age.
3. Willingness to donate gingival tissue and collect a microbiological sample for the study.

Exclusion criteria:

1. Using systemic antibiotics (intravenous, intramuscular, or oral) in the last six months.
2. Having used corticosteroids or other immunosuppressants (e.g., cyclosporine), cytokine therapy, methotrexate or any other immunosuppressive chemical agent, or high-dose commercially available probiotics (≥ 108 colony-forming units per day) in tablet, capsule, or powder form in the last three months. The use of fermented foods/liquids, e.g., milk, yogurt, etc., does not apply to the exclusion of the individual.
3. Being pregnant or breastfeeding.
4. Subjects who cannot give consent.

Intraoral Examination: All subjects will undergo a full-mouth examination using a specially designed form (Appendix 3). General history (age, biological sex, occupation), habits, diseases, and medications will be recorded. A periodontogram will also be included to record periodontal measurements, probing depths, clinical attachment loss, bleeding on probing, etc.

Sample Collection: Representative gingival collar biopsies (2 mm wide) will be collected under local anesthesia and placed in 4% formalin for histological analysis, T-PER (Thermofisher Scientific) for Western blot analysis, and RNA later (Thermofisher Scientific) for RT-qPCR analysis. In healthy subjects, these samples will be collected as biological waste and may be obtained, for example, in the following cases: crown lengthening surgeries, third molar extractions, or teeth where there is no significant risk of removing gingival tissue, molar areas with opercula, or gingiva covering part of the dental crown where removing gingival tissue is not a risk. In subjects with periodontitis and peri-implantitis, these samples will be collected during procedures before subgingival instrumentation and/or periodontal or peri-implant surgery in the most affected area at probing depths.

1. STAT3 activation in gingival tissue during gingival health, periodontitis, and peri-implantitis: For samples stored in T-PER, protein extraction will be performed, and total STAT3 and its activation (pSTAT3) will be determined using Western blot using antibodies that recognize STAT3 and pSTAT3 at Tyr705 (Cell Signaling Technology, USA). GAPDH will be used as a loading control, and the bands obtained will be quantified using ImageJ software (NIH, Bethesda, USA).
2. Characterization of pSTAT3 in gingival tissue during gingival health, periodontitis, and peri-implantitis: For samples fixed in 4% formalin, the localization of pSTAT3 (epithelium and connective tissue) will be determined using immunofluorescence using antibodies that recognize CD45 for immune cells, Ck5 for epithelial cells, and pSTAT3 for the activated protein. The co-localization of pSTAT3-Ck5 and pSTAT3-CD45 will be determined by confocal microscopy at 40x.
3. Analysis of the pSTAT3-mediated immune-defense response in gingival tissue during gingival health, periodontitis, and peri-implantitis: For samples stored in RNA later, total RNA will be extracted, and the following genes associated with the immune-defense response will be amplified using the RT-qPCR technique:

ELIGIBILITY:
Inclusion Criteria:

Patients in the gingival health group:

1. Meet the case definition of gingival health (Chapple et al. 2018).
2. ≥ 18 years of age.
3. Willingness to donate gingival tissue and collect microbiological samples for the study.

Patients in the periodontitis group:

1. Meet the case definition of periodontitis (Papapanou et al. 2018).
2. ≥ 18 years of age.
3. Willingness to donate gingival tissue and collect microbiological samples for the study.

Patients in the peri-implantitis group:

1. Meet the case definition of periodontitis and peri-implantitis (Berglundh et al., 2018).
2. ≥ 18 years of age.
3. Willingness to donate gingival tissue and collect a microbiological sample for the study.

Exclusion Criteria

- 1. Having used systemic antibiotics (intravenous, intramuscular, or oral) in the last six months.

2. Having used corticosteroids or other immunosuppressants (e.g., cyclosporine), cytokine therapy, methotrexate, or any other immunosuppressive chemical agent, or high-dose commercially available probiotics (≥ 108 colony-forming units per day) in tablet, capsule, or powder form within the last three months. The use of fermented foods/liquids, e.g., milk, yogurt, etc., does not apply to the exclusion of the individual.

3. Being pregnant or breastfeeding. 4. Subjects who cannot give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects over 17 years of age who attend the Dental Clinic of the Faculty of Dentistry of the University of Chile and present with a diagnosis of gingival health, periodontitis, and peri-implantitis, according to the classification of periodontal and peri-implant diseases (Caton et al., 2018), will be recruited and examined.
  All subjects must sign an informed consent form previously validated by an ethics committee and meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Percentage of epithelial cells that present activated STAT3 protein | Baseline
  Measured as a percentage of epithelial cells that present the activated protein from 0 to 100, where 0 means no epithelial cells activate the protein, and 100% means all cells present it.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No